CLINICAL TRIAL: NCT01907724
Title: A Phase I, Randomized, Multiple-Dose Study to Evaluate the Pharmacokinetic Drug-Drug Interaction Between IDX719, Simeprevir, TMC647055 and Ritonavir When Administered in Combination in Healthy Subjects
Brief Title: Drug-Drug Interaction Between IDX719, Simeprevir, TMC647055 and Ritonavir When Administered in Combination in Healthy Participants (MK-1894-007)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1894-007; IDX-06A-007 (Other: Idenix Protocol Number)
Record Dates: First submitted 2013-06-04; First posted 2013-07-25 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Hepatitis C, Chronic
Keywords: Chronic hepatitis C; Hepatitis C virus; HCV
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — samatasvir; Simeprevir; 27-cyclohexyl-12,13,16,17-tetrahydro-22-methoxy-11,17-dimethyl-10,10-dioxide-2,19-methano-3,7:4,1-dimetheno-1H,11H-14,10,2,9,11,17-benzoxathiatetraazacyclo docosine-8,18(9H,15H)-dione; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDX719 + RTV (Experimental): Participants take IDX719 150 mg once daily (QD) + ritonavir 30 mg QD on Days 1-7, and then take IDX719 150 mg QD + simeprevir 75 mg QD + TMC647055 450 mg QD + RTV 30 mg QD on Days 8-14.
  Interventions: Drug: IDX719; Drug: Simeprevir; Drug: TMC647055; Drug: RTV
- Simeprevir/TMC647055 + RTV (Experimental): Participants take simeprevir 75 mg QD + TMC647055 450 mg QD + RTV 30 mg QD on Days 1-7, and then take IDX719 150 mg QD + simeprevir 75 mg QD + TMC647055 450 mg QD + RTV 30 mg QD on Days 8-14.
  Interventions: Drug: IDX719; Drug: Simeprevir; Drug: TMC647055; Drug: RTV

INTERVENTIONS:
Drug: IDX719 — IDX719 will be supplied as a 50 mg tablet for oral administration.
Drug: Simeprevir — Simeprevir will be supplied as 75 mg capsules for oral administration.
  Other Names: Olysio™
Drug: TMC647055 — TMC647055 will be supplied as 150 mg capsules for oral administration.
Drug: RTV — RTV will be supplied as 80 mg/mL solution for oral administration.
  Other Names: Norvir™

SUMMARY:
The purpose of this study is to evaluate the potential for a PK drug-drug interaction when IDX719, simeprevir, TMC647055 and low-dose ritonavir (RTV) are administered in combination. Safety and tolerability will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Agrees to use a double method of birth control (one of which must be a barrier) from Screening through at least 90 days after the last dose of the study drug
* Male participants agree not to donate sperm from Day -1 through 90 days after the last dose of study drug

Exclusion Criteria:

* Is pregnant or breastfeeding
* Has another clinically significant medical conditions or laboratory abnormality(s)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Observed maximum plasma drug concentration (Cmax) | Up to 14 days
Time to maximum concentration (Tmax) | Up to 14 days
Area under the drug concentration-plasma time curve from time zero to last measurable concentration (AUC0-t) | Up to 14 days
Predose trough concentration (Ctrough) | Up to 14 days
Apparent terminal elimination rate constant | Up to 14 days
Observed terminal half-life (T1/2) | Up to 14 days

SECONDARY OUTCOMES:
Percentage of participants experiencing serious adverse events (SAEs) | Up to 28 days
Percentage of participants experiencing adverse events (AEs) | Up to 28 days
Percentage of participants with Grade 1-4 laboratory abnormalities | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC